CLINICAL TRIAL: NCT03056326
Title: A Phase I, Randomised, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of Inhaled CHF 6333 After Single and Repeated Ascending Doses in Healthy Male Subjects
Brief Title: A Study to Investigate Safety, Tolerability and Pharmacokinetics of Single and Repeat Doses of CHF6333 in Healthy Subjects
Acronym: CHF6333 FIH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-06333AA1-01; 2015-005552-94 (EudraCT Number)
Record Dates: First submitted 2017-02-03; First posted 2017-02-17 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Non-Cystic Fibrosis Bronchiectasis; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Part 1: alternating cross-over design
  Part 2: parallel design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHF6333 Active (Experimental)
  Interventions: Drug: CHF6333 (Part 1 - SAD); Drug: CHF6333 (Part 2 - MAD)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (Part 1 - SAD); Drug: Placebo (Part 2 - MAD)

INTERVENTIONS:
Drug: CHF6333 (Part 1 - SAD) — Single doses of CHF6333 at each period
  Arms: CHF6333 Active
Drug: Placebo (Part 1 - SAD) — Single doses of placebo matching CHF6333 at each period
  Arms: Placebo
Drug: CHF6333 (Part 2 - MAD) — once daily multiple doses of CHF6333 for 14 days
  Arms: CHF6333 Active
Drug: Placebo (Part 2 - MAD) — once daily multiple doses of placebo matching CHF6333 for 14 days
  Arms: Placebo

SUMMARY:
Human Neutrophil Elastase (HNE) plays a pivotal role in innate immunity and in neutrophilic lung inflammation that characterized many diseases. CHF 6333 is a potent and 24h-durable inhibitor of HNE, developed as Dry Powder Inhaler (DPI) formulation. This study is designed to investigate the tolerability, safety and pharmacokinetics of inhaled CHF6333 DPI in healthy male subjects.

The study will comprise two parts:

Part 1 will consist of two alternated cohorts of healthy male subjects to assess the safety, tolerability and pharmacokinetics of Single Ascending Dose (SAD) of CHF6333.

Part 2 will consist of four sequential cohorts of healthy male subjects to assess the safety, tolerability and pharmacokinetics of Multiple Ascending Dose (MAD) of CHF6333

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged 18-55 years
* BMI between 18-30 kg/m2
* Non smokers
* Lung function above 80% of predicted normal value
* Healthy subjects based on medical evaluation including medical history, physical examination, laboratory tests and cardiac testing

Exclusion Criteria:

* Any clinically relevant abnormalities and/or uncontrolled diseases
* Abnormal laboratory values
* Recent respiratory tract infection
* Hypersensitivity to the drug or excipients
* Positive serology results
* Positive cotinine, alcohol, drug of abuse tests
* Unsuitable veins for repeated venepuncture

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2016-11; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Adverse events | Part 1 from Day 1 to 5, Part 2 from Day 1 to 15
  Treatment-related Adverse events
Change in Vital signs | Part 1 from Day 1 to 5, Part 2 from Day 1 to 15
  Blood pressure
Heart Rate | Part 1 Day 1-2, Part 2 Day 1-2 and Day 14-15
  Change in Heart Rate (from ECG)
QTcF interval | Part 1 Day 1-2, Part 2 Day 1-2 and Day 14-15
  Change in QTcF interval (from ECG)
PR interval | Part 1 Day 1-2, Part 2 Day 1-2 and Day 14-15
  Change in PR interval (from ECG)
QRS interval | Part 1 Day 1-2, Part 2 Day 1-2 and Day 14-15
  Change in QRS interval (from ECG)
Holter recording abnormalities | Part 1 Day 1-2, Part 2 Day 1-2 and Day 14-15
  24h-holter ECG recording
FEV1 | Part 1 Day 1-2, Part 2 Day 1-14-15
  Change in FEV1 (Forced exhalation volume in the first second)
Clinical chemistry and haematology | Part 1 Day 1-5, Part 2 Day 1-15
  change in Clinical chemistry and haematology parameters
Urinalysis | Part 1 Day 1-5, Part 2 Day 1-15
  Change in urinalysis parameters

SECONDARY OUTCOMES:
Area under the plasma concentration | Part 1 from Day 1 to 5, Part 2 from Day 1-2 and Day 14-15
Peak plasma concentration (Cmax) | Part 1 from Day 1 to 5, Part 2 from Day 1-2 and Day 14-15
  maximum plasma concentration of CHF6333
Time to reach the maximum plasma concentration (tmax) | Part 1 from Day 1 to 5, Part 2 from Day 1-2 and Day 14-15
Elimination half-life (t1/2) | Part 1 from Day 1 to 5, Part 2 from Day 1-2 and Day 14-15
Clearance (CL/F) | Part 1 from Day 1 to 5, Part 2 from Day 1-2 and Day 14-15
  Absolute plasma clearance
Volume of distribution (Vz/F) | Part 1 from Day 1 to 5, Part 2 from Day 1-2 and Day 14-15
  plasma volume of distribution
Urinary excretion (Ae) | Part 1 from Day 1 to 5, Part 2 from Day 1-2 and Day 14-15
  Amount of CHF6333 excreted in urine
fraction excreted (fe) | Part 1 from Day 1 to 5, Part 2 from Day 1-2 and Day 14-15
  Percentage of drug excreted in urine
Renal clearance (CLr) | Part 1 from Day 1 to 5, Part 2 from Day 1-2 and Day 14-15

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, Principal Investigator — SGS Life Sciences, a division of SGS Belgium NV
Locations (1):
- SGS Life Sciences, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided